CLINICAL TRIAL: NCT06679621
Title: A Telehealth Intervention to Increase Patient Preparedness for Surgery in Latinas
Acronym: TIPPS-Urogyn
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Gabriela Halder, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 300012104; 1K23HD115269 (NIH)
Record Dates: First submitted 2024-11-05; First posted 2024-11-07 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Incontinence; Prolapse
MeSH Terms: conditions — Prolapse

STUDY DESIGN:
Intervention Model Description: The randomized design is for Aim 3 of our study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Routine Preoperative Counseling (No Intervention): Participants scheduled to undergo urogynecologic surgery will receive routine preoperative counseling.
- Telehealth intervention (Experimental): Patient scheduled to undergo urogynecologic surgery will receive routine preoperative counseling in addition to the modified telehealth intervention.
  Interventions: Behavioral: Telehealth intervention

INTERVENTIONS:
Behavioral: Telehealth intervention — This telehealth intervention will be made using human centered design methods
  Arms: Telehealth intervention

SUMMARY:
There are 3 aims of this study. In Aim 1 community patient partners will be enrolled to help guide the research being performed in all of the aims. Investigators will also administer a survey that will help determine factors associated with surgical preparedness. In Aim 2 investigators will develop an intervention to increase surgical preparedness using Human Centered Design Methods. Aim 3 will pilot test the intervention using mixed methods to determine feasibility and implementation outcomes.

DETAILED DESCRIPTION:
The purpose of this project is to understand surgical preparedness in Latinas undergoing urogynecologic surgery and to develop TIPPS-Latina a refined version of our telehealth intervention for Latinas undergoing urogynecologic surgery using HCD and D&I methods. The goal of the first aim is to develop a participatory design approach and understand surgical preparedness in Latinas undergoing urogynecologic surgery. This cross-sectional study will run in parallel to the other aims. The participatory action framework will guide Aims 1-3. The goals of Aim 2 and Aim 3 are develop and test TIPPS-Latina using the Discover, Design/Build, and Test (DDBT) framework, which is a HCD method to generate evidence-based interventions and their implementations9. During the Discover phase investigators will identify preferences for refinement of TIPPS-Latina and its contextual deployment using mixed methods. During the Design/Build phase investigators will use an iterative process to generate, modify, and adapt our intervention. During the Test phase investigators will conduct pilot testing of TIPPS-Latina using a mixed methods approach that determines feasibility and implementation outcomes. Throughout our study, surgical preparedness will be measured using the Surgical Preparedness Assessment (SPA), a validated survey for measuring preparedness in women undergoing urogynecologic surgery that was developed by our group

ELIGIBILITY:
Inclusion Criteria:

Patients who

* Self-report as female
* 18 years and older
* Self-report as Hispanic ethnicity
* Scheduled to undergo a surgery for a urogynecologic condition in the operating room (surgery to correct pelvic organ prolapse, urinary/fecal incontinence, fistula, urethral masses)
* Able to read and write English and/or Spanish

Urogynecologists who -Routinely perform urogynecologist surgeries to correct pelvic organ prolapse, urinary/fecal incontinence, fistula, urethral masses

Nurses who

* Spend most of their time at a urogynecologic clinic
* Engage in the process of preparing patients for urogynecologic surgery

Exclusion Criteria:

Patients who

* Self-report as male
* Are less than 18 years of age
* Self-report as not of Hispanic ethnicity
* Scheduled to undergo a surgery for a condition that is not urogynecologic or is not in the operating room
* Patients undergoing procedures that are traditionally performed in the office (bladder Botox, pelvic floor Botox, urethral bulking)

Urogynecologists who

-Do not routinely perform urogynecologic surgery

Nurses who

* Do not spend most of their time at a urogynecology clinic
* Do not engage in the process of preparing patients for urogynecologic surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 357 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the Intervention | Day of Surgery, before surgery, in the preoperative holding
  A feasible study will be defined a 1) >4 on 1-5 Likert-type scales of acceptability, appropriateness, and feasibility; 2) >70% for adherence; and 3)> 90% for dose delivery, and percent completed intervention.
  Acceptability will be measured by the Acceptability of the Intervention Measure Appropriateness will be measured by the Intervention Appropriateness Measure Feasibility will be measured by the Feasibility of Intervention Measure
Acceptability of the Intervention | Day of Surgery, before surgery, in the preoperative holding
  As measured by the Acceptability of the Intervention Measure
Appropriateness of the Intervention | Day of Surgery, before surgery, in the preoperative holding
  As measured by the Intervention Appropriateness Measure

SECONDARY OUTCOMES:
Surgical Preparedness | Day of Surgery, before surgery, in the preoperative holding
  As measured by the Surgical Preparedness Assessment survey
Health Literacy | Preoperative Visit, before surgery
  As measured by the Brief Health Literacy Screen
Self-Efficacy | Preoperative Visit, before surgery
  As measured by the General Self-Efficacy Scale
Trust in Provider | Preoperative Visit, before surgery
  As measured by the Trust in Provider Scale
Decisional Conflict | Day of Surgery, before surgery, in the preoperative holding
  As measured by the Decisional Conflict Scale
Postoperative Anxiety/Depression | Preoperative Visit, before surgery
  As measured by the Hospital Anxiety/Depression Scale
Satisfaction with Healthcare Services | Postoperative Visit 6-8 weeks after surgery
  As measured by the CAHPS Clinician & Group Visit Adult Survey

OTHER OUTCOMES:
Demographics | Preoperative Visit 6-8 weeks after surgery
  Baseline Case Report Form
Surgical Data | Day of Surgery, before surgery, in the preoperative holding
  Surgical Case Report Form
Adverse Events | Postoperative Visit 6-8 weeks after surgery
  Adverse Events Case Report Form
Symptom Bother - PFDI 20 | Preoperative Visit, before surgery and Postoperative Visit 6-8 weeks after surgery
  As measured by the Pelvic Floor Distress Inventory-20
Symptom Bother - PGI-S | Preoperative Visit, before surgery and Postoperative Visit 6-8 weeks after surgery
  As measured by the Global Impressions of Severity
General Health | Preoperative Visit, before surgery and Postoperative Visit 6-8 after surgery
  EQ-5D-5L
Self-Esteem | Preoperative Visit, before surgery
  Rosenberg Self-Esteem Scale

CONTACTS AND LOCATIONS:
Overall Officials: Gabriela Halder, MD, MPH, Principal Investigator — Assistant Professor
Locations (1):
- University of Alabama Birmginham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No